CLINICAL TRIAL: NCT01458041
Title: Iloprost Therapy in Patients With Critical Limb Ischemia: Evaluation of Efficacy and Safety
Brief Title: Iloprost Therapy in Patients With Critical Limb Ischemia
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 15439; VE1011HU (Other: Company Internal)
Record Dates: First submitted 2011-10-10; First posted 2011-10-24 (Estimated); Last update posted 2015-03-02 (Estimated); Status verified 2015-02

CONDITIONS: Peripheral Arterial Disease
Keywords: Critical limb ischaemia; Iloprost; Quality of life; Visual analogue scale
MeSH Terms: conditions — Peripheral Arterial Disease; Chronic Limb-Threatening Ischemia | interventions — Iloprost

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Group 1
  Interventions: Drug: Iloprost (Ilomedin, BAYQ6256)

INTERVENTIONS:
Drug: Iloprost (Ilomedin, BAYQ6256) — Prescription and treatment of Iloprost will be decided by physicians

SUMMARY:
Monitoring efficacy and safety aspects of iv. iloprost therapy of patients with critical limb ischemia by recording clinical parameters.

ELIGIBILITY:
Inclusion Criteria:

* Patients who fulfill the internationally defined criteria of critical limb ischemia;
* Patients who are not eligible for vascular surgery or angioplasty interventions and
* Patients who are treated with iloprost infusion.
* The treating physician has decided iloprost treatment before study enrollment.

Exclusion Criteria:

* Exclusion criteria are in accordance with the Summary of Product Characteristics of Ilomedin.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hospitalized patients
Sampling Method: Non-Probability Sample
Enrollment: 126 (Actual)
Dates: Start 2011-08; Primary Completion 2014-05 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Change of limb pain at rest assessed by visual analogue scale | At baseline, at the end of iloprost treatment, at follow-up visits ( month 3, 6, 12)
  Pain relief will be defined as complete relief of pain while off analgesics

SECONDARY OUTCOMES:
Incidence of ulcer healing | at baseline, at the end of iloprost treatment and at follow-up visits ( month 3, 6, 12)
Collection of interventional / surgical procedures including 1) Rate of revascularization procedures; 2) Minor amputations; 3) Frequency and height of major amputations | at baseline, at the end of iloprost treatment and at follow-up visits ( month 3, 6, 12)
Mortality and/or severe cardiovascular events (AMI, stroke) | at baseline, at the end of iloprost treatment and at follow-up visits ( month 3, 6, 12)
Hemodynamic measurements: peripheral arterial blood flow and pressure on ankle / hallux level by Doppler scanner | at baseline, at the end of iloprost treatment and at follow-up visits ( month 3, 6, 12)
Changes of transcutaneously measured tissue oxygen tension values | at baseline, at the end of iloprost treatment and at follow-up visits ( month 3, 6, 12)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Many Locations, Hungary